CLINICAL TRIAL: NCT06886360
Title: An Open-label Study of Patients with Primary Sclerosing Cholangitis (PSC) Treated with Norucholic Acid Tablets
Brief Title: Study with Norucholic Acid Tablets in Patients with Primary Sclerosing Cholangitis (PSC)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NUT-022/PSC; 2024-514292-18-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- norucholic acid 1500 mg/day (Experimental): 3 film-coated tablets once daily for 72 weeks containing in total norUrsodeoxycholic acid 1500 mg
  Interventions: Drug: norucholic acid

INTERVENTIONS:
Drug: norucholic acid — 500 mg norucholic acid film-coated tablets; 3 tablets/day

SUMMARY:
Open-label, multi-center, phase III trial. Oral treatment with 1500 mg norucholic acid in Primary Sclerosing cholangitis

ELIGIBILITY:
Inclusion criteria:

1. Signed informed consent.
2. Males or females ≥ 18 years.
3. Patient has previously been diagnosed with PSC, has participated in the previous NUC 5/PSC trial and has completed the DBE phase with Visit 22, or has prematurely terminated the DBE phase before this trial has been started, or has prematurely terminated the DBE phase after this trial has been started, under the condition that the premature termination was due to lack of efficacy*. (*Lack of efficacy as defined in the NUC-5/PSC trial.)

Exclusion Criteria:

1. History or presence of chronic alcoholic consumption (daily consumption > 30 g in men, > 20 g in women).
2. Patients who discontinued study participation in NUC-5/PSC due to an AE possibly caused by the study drug.
3. Liver Cirrhosis or any cirrhosis-related symptoms which in the opinion of the investigator may affect the patient's safety.
4. History of liver transplantation or patient listed for transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment emergent adverse events | 72 weeks from enrollment to end of treatment
Occurrence of serious treatment emergent adverse events | 72 weeks from enrollment to end of treatment
Occurrence of severe treatment emergent adverse events | 72 weeks from enrollment to end of treatment
Occurrence of adverse drug reactions | 72 weeks from enrollment to end of treatment
Occurrence of unexpected treatment emergent adverse events | 72 weeks from enrollment to end of treatment
Occurrence of treatment emergent adverse events leading to study withdrawal | 72 weeks from enrollment to end of treatment
Occurrence of adverse events leading to death | 72 weeks from enrollment to end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Trauner, MD, Principal Investigator — Medical University of Vienna, dept. of Internal Medicine III

IPD SHARING:
Plan to Share IPD: No
It is not decided which data will be made available. A time frame cannot be indicated yet.